CLINICAL TRIAL: NCT00603824
Title: Fondaparinux in Patients With Acute Heparin-Induced Thrombocytopenia
Brief Title: Fondaparinux in Patients With Acute Heparin-Induced Thrombocytopenia (HIT)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PI relocated
Sponsor: Methodist Healthcare (Other)
Collaborators: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MHIRB # 2007-058
Record Dates: First submitted 2008-01-04; First posted 2008-01-29 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2009-06

CONDITIONS: Heparin-Induced Thrombocytopenia
Keywords: heparin-Induced thrombocytopenia; fondaparinux
MeSH Terms: interventions — Fondaparinux; argatroban; lepirudin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Fondaparinux
  Interventions: Drug: fondaparinux
- B (Active Comparator): Direct thrombin inhibitor
  Interventions: Drug: argatroban or lepirudin

INTERVENTIONS:
Drug: fondaparinux — fondaparinux subcutaneous injection once daily until INR stable in therapeutic range, at least five days: 5 mg if less than 50 kg, 7.5 mg if 50-100 kg, 10 mg if >100 kg
  Other Names: Arixtra
  Arms: A
Drug: argatroban or lepirudin — continuous infusion titrated into therapeutic range and for at least 5 days and until INR stable in therapeutic range
  Other Names: Refludan
  Arms: B

SUMMARY:
The purpose of this study is to test the safety and efficacy of fondaparinux in patients with heparin-induced thrombocytopenia (HIT). The primary objective is to ensure that patients with HIT who are treated with fondaparinux experience a prompt and complete recovery of their platelet count, and the secondary objective is to determine if any new blood clots are formed while receiving the fondaparinux and up to one month after study enrollment. This information will be compared to a historical control.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age;
* If female of childbearing potential, negative pregnancy test result;
* Diagnosis of HIT confirmed by the following: Decreased platelet count by 50% or greater OR platelets < 100,000/mm3 during or within 2 weeks after heparin exposure and/or new thromboembolic complications during or within 2 weeks after heparin exposure;
* Laboratory confirmation (either heparin PF4 antibody or serotonin release assay positive).

Exclusion Criteria:

* Estimated creatinine clearance less than 30 ml/min (either measured or by using Cockcroft Gault equation);
* Pregnancy or lactating;
* Blood dyscrasia other than HIT;
* History of thrombocytopenia associated with fondaparinux;
* Recent (within 6 weeks) or planned surgery of CNS, eye or traumatic surgery resulting in large open surfaces or other procedures with high bleeding risk or if lumbar puncture is planned;
* Active bleeding of GI tract, GU tract, CNS or respiratory tract;
* Malignant hypertension, pericarditis, pericardial effusion, endocarditis or eclampsia;
* Inadequate laboratory facilities, inadequate support system at home, alcoholism, drug abuse, psychosis or dementia;
* Hypersensitivity or contraindication to warfarin or fondaparinux.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2009-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Platelet count recovery | 5 days

SECONDARY OUTCOMES:
Recurrent thromboembolic complications | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bob L Lobo, Pharm.D., Principal Investigator — Methodist University Hospital; Sohail Minhas, MD, Principal Investigator — University of Tennessee